CLINICAL TRIAL: NCT05478447
Title: Effect of Sympathetic Stress on Whole Body Vibration Reflex
Brief Title: Sympathetic Stress and Whole Body Vibration Reflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan KARACAN, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SSTWBVR
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Vibration; Exposure; Muscle Physiology
Keywords: tonic vibration reflex; vibration; whole body vibration; sympathetic activation
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibration group (Experimental): Vibration (WBV, and tendon vibration) and sympathetic activation maneuvers will be applied to participants
  Interventions: Procedure: Vibration

INTERVENTIONS:
Procedure: Vibration — whole-body vibration, and tendon vibrations will be applied to the human body
  Other Names: whole body vibration; tendon vibration; sympathetic activation maneuver

SUMMARY:
Whole body vibration (WBV) is a therapeutic modality in the form of exercise on a vibrating platform with an amplitude of 2-4 mm at a frequency of 25-50 Hz, which is used with increased popularity in sports medicine and rehabilitation due to its beneficial effects on muscle strength, balance, postural control, bone formation, and circulation. Beneficial effects on muscle strength and athletic performance have been reported. Spinal reflexes explain these beneficial neuromuscular effects. However, the neuronal circuit and receptors of the reflex response have not been defined precisely. A group of researchers propose that the reflex system underlying the neuromuscular effects of WBV is the Tonic vibration reflex (TVR), whose receptor is the muscle spindle; other researchers claim that the reflex latency induced by WBV is 4-5 ms longer than the TVR latency, so it is a bone myoregulation reflex whose receptor is osteocytes.

The muscle spindle has sympathetic innervation. It has been reported that in case of increased sympathetic activity, muscle spindle sensitivity may increase and short-latency stretch reflex may be facilitated. The variation of muscle spindle activity with sympathetic activity may provide an opportunity to define the nature of the reflex response during WBV. Muscle spindles are more sensitive to vibrations around 100 Hz. This study has two hypotheses: According to the first hypothesis, WBV activates muscle spindles and the reflex latency induced by WBV is the same as TVR latency, and the latency does not change with increased sympathetic activity. According to the alternative hypothesis, WBV activates osteocytes, and WBV-induced reflex latency is longer than TVR latency. With increased sympathetic activity, the WBV reflex becomes dominant and the WBV-induced reflex latency becomes shorter. The aim of this research is to determine which of these two hypotheses is valid.

DETAILED DESCRIPTION:
22 healthy males between the ages of 20 and 45 will be recruited for this study. All subjects will receive pre-study informed consent. All experimental procedures were designed with the Helsinki declaration in mind and approved by the local ethics committee. In all subjects, whole body vibration(WBV) and isolated tendon vibration will be applied before, after, and during sympathetic activation maneuvers. Reflex responses induced by WBV and isolated tendon vibration will be recorded by surface electromyography (EMG) from the right soleus muscle. Latency calculation will be made using the "Cumulative averaging method".

Mental arithmetic task and cold stress test will be applied as sympathetic activation maneuver. For the mental arithmetic task, the subject is asked to mentally subtract a two-digit number from a four-digit number and respond within five seconds. This arithmetic calculation is repeated for different numbers. This test is continued for two minutes. For the cold stimulation test, subjects are asked to dip their right hand into 2-4 degrees cold water up to the elbow and hold it in the water for two minutes. At this time, either WBV or tendon vibration will be applied. After a ten-minute break, a cold stimulation test will be applied to the left hand and the subject will be asked to do mental arithmetic calculations simultaneously. Meanwhile, other vibrations will be used. The sympathetic response will be evaluated by heart rate and sympathetic skin response.

Whole body vibration will be applied to the right leg while subjects are sitting with their knee, hip, and ankle joints in a 90-degree position.

The left leg will rest on a vibration-isolated platform. During this position, he will be asked not to voluntarily contract the calf muscle. The vibration will be applied with the PowerPlate® Pro5 WBV (London UK) device. The vibration amplitude will be 2.2 mm. The vibration frequency will be 30, 35, 40, and 45 Hz. Each vibration frequency will be applied for 30 seconds. A 5-second rest period will be applied between 30-second vibrations. Piezo-electric accelerometer (LIS344ALH, full-scale of ± 6 g, linear accelerometer, ECOPACK®, Mansfield, TX, USA) will be fixed on the WBV device platform for reflex latency calculation. For tonic vibration 100, 135, 150, and 180 Hz vibrations will be applied to the Achilles tendon. 30 seconds of vibration will be applied at each frequency. A direct current (DC) motor vibrator will be used to apply this vibration (Bosch™, amplitude 2 mm, motor speed 5000-20000 / min). A piezo-electric accelerometer (LIS344ALH, full-scale of ± 6 g, linear accelerometer, ECOPACK®, Mansfield, TX, USA) will be placed on the skin of the Achilles tendon to calculate the tonic vibration reflex latency. Superficial EMG recordings will be taken from the right soleus muscle with the bipolar technique. A pair of self-adhesive Ag/AgCl (KENDALL® Coviden, Massachusetts, USA) electrodes will be attached to the skin. The electrodes on the soleus will be positioned according to the SENIAM protocol. The ground electrode will have adhered to the right lateral malleolus. Before the electrodes are attached to the skin, if there are hairs on the skin, they will be shaved and the oil layer on the skin will be cleaned with alcohol cotton. In order to increase the moisture of the skin, ECG gel will be applied to the skin area where the electrode will be attached. Superficial EMG recordings will be taken with a PowerLab ® (ADInstrument ADInstruments, Oxford, UK) data recorder with a sample rate of 40 kHz.

EMG recordings will be analyzed offline with LabChart7 Pro® version 7.3.8 (ADInstrument, Oxford, UK). The acceleration measurement data will be recorded with the PowerLab (ADInstrument London) data logger simultaneously with the EMG recording. Acceleration recording will be made with a sample rate of 40 kHz. Simultaneously, heart rate and sympathetic skin response will be captured with a Biopac (Biopac System Inc CA) data recorder at a rate of 20 kHz.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Being a young adult (20-45 years old)
* Volunteer
* Male

Exclusion Criteria:

* Scar, dermatitis, etc. in the skin tissue where EMG electrodes will be placed
* Kidney stone history
* Fracture in the lower extremity, history of orthopedic surgery
* Heart disease, Hypertension
* Dizziness
* Metabolic bone diseases, including osteoporosis
* History of bone occupying lesion, neoplasia, osteomyelitis
* Degenerative, inflammatory diseases of the joints of the lower extremities
* Lower extremity thrombophlebitis
* Lower extremity motor loss, sensory loss, muscle atrophy
* Cold allergy
* Subjects who cannot tolerate whole-body vibration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Whole-body vibration (WBV) induced reflex latency | during intervention, an average of 3 minute
  Latency of the soleus reflex response induced by WBV. Its unit is milliseconds
Tendon vibration induced reflex latency | during intervention, an average of 3 minute
  Vibration will be applied to the achilles tendon. The soleus reflex latency induced by the tendon vibration will be measured. Its unit is milliseconds

SECONDARY OUTCOMES:
Heart rate variability | during intervention, an average of 2 hours
  Heart rate variability will be measured to determine sympathetic activity. Low-frequency (LF) and high-frequency (HF) were considered to reflect sympathetic and parasympathetic activity, respectively. The autonomic balance was obtained by the ratio between the sympathetic and parasympathetic areas (LF/HF); wherein ratios >1, <1, and 1 were indicative of sympatheticotonia, vagotonia, and sympathovagal balance, respectively.
Sympathetic skin response | during intervention, an average of 2 hours
  Sympathetic skin response will be measured to determine sympathetic activity.Unit is milliVolt

CONTACTS AND LOCATIONS:
Overall Officials: İlhan Karacan, Assoc Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)